CLINICAL TRIAL: NCT01086774
Title: Efficacy of Systane Balance to Stabilize the Tear Film in Dry Eye Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-09-39
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry eye; Tear Film Stability
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Systane Ultra (Experimental): Systane Ultra Lubricant Eye Drops
  Interventions: Other: Systane Ultra Lubricant Eye Drops

INTERVENTIONS:
Other: Systane Ultra Lubricant Eye Drops — Single drop in both eyes

SUMMARY:
Evaluation of the optical effects of Systane Ultra

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. Subjects must have Tear Break Up Time (TBUT) < 5 seconds
3. Subjects must have a maximum blink interval (MBI) < 10 seconds
4. Subjects must be willing to comply with all study requirements.
5. Subjects must understand, sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

1. Subjects for whom both eyes do not meet all inclusion criteria and either eye meets exclusion criteria
2. Subjects who are pregnant, lactating or planning to be pregnant during the course of the study
3. Subjects with known sensitivity to planned study concomitant medications
4. Subjects participating in any other ophthalmic drug or device clinical trial within 30 days of this clinical investigation.
5. Use of ocular drugs, other than study medications, during the study and within 14 days prior to study entry or any other ocular medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Improvement in maximum blink interval (MBI) | 1 day

SECONDARY OUTCOMES:
Tear film stability and contrast sensitivity | 1 day